CLINICAL TRIAL: NCT02580370
Title: Safety and Efficacy of Botulinum Toxin Type A Topical Gel for Lateral Canthal Lines
Acronym: REALISE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RT001-CL038
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Skin Aging
Keywords: REALISE 1
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose A (Experimental): Botulinum toxin type A
  Interventions: Biological: Botulinum toxin type A
- Dose B (Placebo Comparator): Placebo comparator
  Interventions: Biological: Placebo comparator

INTERVENTIONS:
Biological: Botulinum toxin type A — Topical botulinum toxin type A
  Arms: Dose A
Biological: Placebo comparator — Topical placebo comparator
  Arms: Dose B

SUMMARY:
This is a safety and efficacy study of botulinum toxin type A in subjects with lateral canthal lines.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Moderate to severe lateral canthal lines when evaluated at rest based on the investigator's global assessment
* Moderate to severe lateral canthal lines when evaluated at rest based on the patient assessment of severity

Exclusion Criteria:

* Any neurological condition that may place the subject at increased risk with exposure to botulinum toxin type A such as amyotrophic lateral sclerosis and motor neuropathy, Lambert-Eaton syndrome, and myasthenia gravis
* Muscle weakness or paralysis, particularly in the area receiving study treatment
* Active skin disease or irritation or disrupted barrier at the treatment area
* Active eye disease or irritation
* Eyelid ptosis, excessive dermatochalasis, deep dermal scarring, or inability to substantially effect the LCL to be treated by manually spreading the skin apart
* Use of topical prescription retinoid product(s) in the lateral canthal areas during the 3 months prior to Screening
* Undergone any procedures that may affect the lateral canthal region during the 12 months prior to Screening
* Treatment with botulinum toxin type A in the lateral canthal areas in the 6 months prior to Screening or 3 months anywhere else in the body

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Composite endpoint based upon the investigator global assessment (IGA-LCL) and patient assessment of severity (PSA) of lateral canthal lines | Week 4

SECONDARY OUTCOMES:
Investigator Global Assessment with 2 points or greater improvement from baseline | Week 4
  Proportion of subjects with 2 points or greater improvement from baseline using the Investigator Global Assessment
Investigator Global Assessment with 1 point or greater improvement from baseline | Week 4
  Proportion of subjects with 1 point or greater improvement from baseline using the Investigator Global Assessment
Patient Severity Assessment with 2 points or greater improvement from baseline | Week 4
  Proportion of subjects with a 2 point or greater improvement from baseline using the Patient Severity Assessment
Patient Severity Assessment with 1 points or greater improvement from baseline | Week 4
  Proportion of subjects with a 1 point or greater improvement from baseline using the Patient Severity Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Coral Gables, Florida, United States